CLINICAL TRIAL: NCT04918134
Title: Investigation on Diagnosis and Treatment of Helicobacter Pylori Infection by Gastroenterologists in Shandong Province
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital, Shandong University
Other Study IDs: 2021-SDU-QILU-G002
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: questionnaire; Helicobacter Pylori Infection; cross-sectional survey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Helicobacter pylori can lead to a variety of digestive system diseases.The eradication of Helicobacter pylori plays an importment role for the treatment of gastrointestinal ulcer and prevention of gastric cancer .Compared with other countries and regions in the world, the infection rate of Helicobacter pylori in China can reach more than 50%. The non-standard diagnosis and treatment of Helicobacter pylori greatly reduces its eradication rate and increases its drug resistance.Therefore, it is very important to strengthen the standardization of diagnosis and treatment to improve the eradication rate.

The purpose of this study is to investigate the diagnosis and treatment status of Helicobacter pylori among gastroenterologists in general hospitals in Shandong Province.It can help us to understand the actual situation of diagnosis and treatment of Helicobacter pylori in hospitals at all levels, and to provide targeted diagnosis and treatment training for doctors.

ELIGIBILITY:
Inclusion Criteria:

* All the gastroenterologists in secondary and tertiary general hospitals of Shandong province

Exclusion Criteria:

* A hospital that does not include gastroenterology
* Hospitals and gastroenterologists that refuse to sign informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Stratified sampling was carried out from all the secondary and tertiary general hospitals in Shandong province, and 120 hospitals were selected.Exclude those without gastroenterology department and those that refused to sign the informed consent, and all gastroenterologists in the hospitals were investigated.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
the results of the questionnaires | 2 months
  the results of each question of the questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hosipital, Jinan, Shandong, China